CLINICAL TRIAL: NCT04502927
Title: Measurements of Displacement Amplitude and Angular Velocities During Passive Extension of the Wrist and Hand Complex in Stroke Patients
Acronym: PHYSIOHAND
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitement issues related to COVID-19
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GHR 1020; IDRCB 2019-A02953-54 (Other: ANSM)
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Muscle Spasticity; Stroke
Keywords: Muscle Spasticity; Mobilization; Wrist and Hand Complex
MeSH Terms: conditions — Muscle Spasticity; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stroke patients with hand spasticity (n=20) (Other)
  Interventions: Procedure: Passive extension mobilization of the hand and wrist joints
- Healthy volunteers (n=10) (Other)
  Interventions: Procedure: Passive extension mobilization of the hand and wrist joints

INTERVENTIONS:
Procedure: Passive extension mobilization of the hand and wrist joints — The physiotherapist will proceed with the passive mobilization of the spastic hand of the stroke patient or the dominant hand for healthy volunteers.
  Two mobilizations will be performed for each participant, i.e. one for each type of medial or lateral grip. The order of mobilization will be determined by randomization.

SUMMARY:
The main objective of this monocentric prospective study is to evaluate the amplitudes and angular velocities of extension of the hand and wrist joints during passive mobilization by a physiotherapist in healthy subjects and stroke patients with spastic hands.

Secondary objectives:

* To compare amplitude and angular velocity values between the group of stroke patients and the group of healthy volunteers,
* To compare amplitude and angular velocity values according to the two types of mobilization (i,e, thumb or fifth finger),
* To assess pain due to mobilization in stroke patients.

DETAILED DESCRIPTION:
Conduct of research:

The realization of the measures will take place at the GHRMSA rehabilitation department.

After receiving the written consent of the study participant, the physiotherapist will proceed with the passive mobilization of the spastic hand of the stroke patient or the dominant hand for healthy volunteers. Videos of the hand will be made using the Darfish system which will allow analysis of the primary endpoint.

Two mobilizations will be performed for each participant, i.e. one for each type of medial or lateral grip. The order of mobilization will be determined by randomization.

ELIGIBILITY:
Eligibility criteria of stroke patients with hand spasticity:

Inclusion Criteria:

* Age ≥ 18 years old
* First stroke diagnosed less than 3 months ago
* Non-functional wrist defined by the Fugl-Meyer Assesment (FMA-EU) upper limb motor subscale with a score ≤45
* Wrist flexor spasticity defined by the Modified Tardieu Scale (MTS) with a rating ≥1
* Written informed consent

Exclusion Criteria:

- None

Eligibility criteria of healthy volunteers:

Inclusion criteria:

* Age ≥ 18 years old
* Written informed consent

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2020-03-18 (Actual)

PRIMARY OUTCOMES:
Amplitude values | 1 minute after intervention
  Amplitude values will be calculated with the Dartfish® system
Angular velocity values | 1 minute after intervention
  Angular velocity values will be calculated with the Dartfish® system

SECONDARY OUTCOMES:
Mean amplitude of the two groups | 1 minute after intervention
Mean angular velocity of the two groups | 1 minute after intervention
Mean amplitude after mobilization with thumb abduction | 1 minute after intervention
Mean angular velocity after mobilization with thumb abduction | 1 minute after intervention
Mean amplitude after mobilization of the fifth finger | 1 minute after intervention
Mean angular velocity after mobilization of the fifth finger | 1 minute after intervention
Pain experienced by stroke patients before mobilisation | 1 minute before intervention
  Pain will be assessed by the Visual Analogue Scale (VAS)
Pain experienced by stroke patients after mobilisation | 1 minute after intervention
  Pain will be assessed by the Visual Analogue Scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Winisdoerffer, Principal Investigator — GHRMSA hospital
Locations (1):
- Groupe Hospitalier de la Région de Mulhouse et Sud Alsace, Mulhouse, France

IPD SHARING:
Plan to Share IPD: No